CLINICAL TRIAL: NCT03006965
Title: Pharmacokinetic Characterization of the Hemophilia A Population in Spain Using an Online Medical Application Based on a Published Population Model and a Bayesian Algorithm
Brief Title: Pharmacokinetic Characterization of the Hemophilia A Population in Spain Using myPKFiT®
Status: Completed | Type: Observational
Sponsor: Spanish Society of Thrombosis and Haemostasis (Other)
Collaborators: Takeda (Industry); Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PK HemoA-SP; STH-OCT-2016-01 (Other: AEMPS)
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Hemophilia A; Hemophilia; Factor VIII Deficiency
Keywords: Hemophilia; Hemophilia A; Factor VIII; Advate; Antithrombotic factor; Pharmacokinetic dosing; Hemarthrosis; myPKFiT
MeSH Terms: conditions — Hemophilia A; Hemarthrosis | interventions — F8 protein, human; Factor VIII; BAX 855

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Whole blood samples collected in citrate plasma tubes to separate it and measure FVIII:chromogenic and FVIII:one stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients: Group of patients in prophylactic treatment with Advate® (octocog alfa) or Adynovi® (rurioctocog alfa pegol), or patients using already myPKFit®.
  Patients will be given a dose of octocog alfa or rurioctocog alfa pegol according to usual clinical practice, and two blood samples will be taken in case of octocog alfa: one sample will be extracted 3-4h postdose (+/- 30 minutes), and the second sample will be extracted 24-32h postdose (+/- 60 minutes). In case of rurioctocog alfa pegol, the first sample is taken in the same conditions than octocog alfa, and the second sample will be extracted 48h postdose (+/- 120 minutes), and other sample post 72h(+/- 120 minutes) optional.
  Interventions: Drug: octocog alfa; Drug: rurioctocog alfa pegol

INTERVENTIONS:
Drug: octocog alfa — Pharmacokinetic Characterization of the Hemophilia A Population in Spain using an standalone web-based software
  Other Names: Advate®; recombinant intravenous factor VIII
Drug: rurioctocog alfa pegol — Pharmacokinetic Characterization of the Hemophilia A Population in Spain using an standalone web-based software
  Other Names: recombinant intravenous factor VIII

SUMMARY:
The purpose of this study is to describe the pharmacokinetic profile of patients with hemophilia A in prophylaxis in Spain using myPKFit®

DETAILED DESCRIPTION:
This pharmacokinetic profile will be obtained in only in patient using Advate® (INN-octocog alfa) or Adynovi® (INN- rurioctocog alfa pegol), both recombinant intravenous FVIII products, with myPKFiT®. This patients will be followed during the period of 12 months, and the pharmacokinetic will be measured collecting at least 2 blood samples, in which the presence of factor VIII will be determined by the usual clinical methods: chromogenic method or coagulative method.

ELIGIBILITY:
Inclusion Criteria:

* Male patients.
* Age between 1 and 65 years old.
* Patients diagnosed with Hemophilia A who are on prophylactic treatment with Advate® or Adynovi® or adjusted with myPKFIT.
* Patients older than 18 who have signed the informed consent form.
* In the case of mature minors, in addition to the consent signed by the legal guardian, an assent of the minor must be obtain.
* In the case of patients legally incapable for giving their consent, their primary caregiver will consent as the patient's legal guardian.

Exclusion Criteria:

* Withdrawal of informed consent.
* Patients with any medical or psychological condition that according to the researcher's criteria prevents them from following the usual clinical practice procedures.
* Patients with concomitant diagnosis of other haemostasis disorders.
* Patients being treated for induction of immunologic tolerance at the time of inclusion.

Ages: 1 Year to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with hemophilia A on prophylactic treatment with Advate® or Adynovi®
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile: FVIII half-life measured with MyPKFiT | 3-4 hours postdose +/- 30 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: FVIII half-life measured with MyPKFiT | 24-32 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: FVIII half-life measured with MyPKFiT | 48 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: FVIII half-life measured with MyPKFiT | 72 hours postdose
  Change from Baseline to 12 months
Pharmacokinetic profile: Clearance measured with MyPKFiT | 3-4 hours postdose +/- 30 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Clearance measured with MyPKFiT | 24-32 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Clearance measured with MyPKFiT | 48 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Clearance measured with MyPKFiT | 72 hours postdose
  Change from Baseline to 12 months
Pharmacokinetic profile: Volume in steady state measured with MyPKFiT | 3-4 hours postdose +/- 30 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Volume in steady state measured with MyPKFiT | 24-32 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Volume in steady state measured with MyPKFiT | 48 hours postdose +/- 60 minutes
  Change from Baseline to 12 months
Pharmacokinetic profile: Volume in steady state measured with MyPKFiT | 72 hours postdose
  Change from Baseline to 12 months

SECONDARY OUTCOMES:
Hemorrhagic risk of physical activity | baseline
  Measured with Broderick scale
Hemorrhagic risk of physical activity | month 12
  Measured with Broderick scale
Joint condition | baseline
  Hemophilia Joint Health Score
Joint condition | month 12
  Hemophilia Joint Health Score
Number of total bleeding episodes in a year | baseline
  Measured by annual bleeding record
Number of total bleeding episodes in a year | month 12
  Measured by annual bleeding record
Annual Joint Bleeding Record | baseline
  Hemophilia Joint Health Score
Annual Joint Bleeding Record | month 12
  Hemophilia Joint Health Score
Self-adherence to treatment evaluation | month 12
  Measured by VERITAS- PRO scale
Adverse Events | baseline
  Collect and identify adverse events
Adverse Events | month 12
  Collect and identify adverse events

CONTACTS AND LOCATIONS:
Overall Officials: M Teresa Álvarez Román, MD,PhD, Principal Investigator — Hospital Universitario La Paz, IdiPAZ, Universidad Autónoma de Madrid
Locations (14):
- Spain (14):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Virgen del Camino, Pamplona, Navarre
  - Hospital Xeral de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Materno-infantil de Málaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided